### Statistical Analysis Plan

| Sponsor | BlackThorn Therapeutics, Inc. |
|---|---|
| Protocol Title: | Phase 2a, Double-blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BTRX-246040 in Parkinson's Disease Subjects with Motor Fluctuations |
| Protocol Number: | NEP-PD-201 |
| Premier Research PCN: | 7311 |
| Document Version: | FINAL Version 1.1 |
| Document Date: | 23-Sep-2019 |





### **Approvals**

| Role | Signatures | Date (dd-Mmm-yyyy) |
|---|---|---|
| Premier<br>Biostatistician | Print Name: Christopher Olson Sign Name: DocuSigned by: christopher ohort Signer Name: christopher olson Signing Reason: I approve this document Signing Time: 22-Nov-2019 15:28:32 EST 4D0BFF36793548808B290E3D71979512 | 22-Nov-2019 15:28:35 Es |
| Premier<br>Biostatistician | Print Name: Adrienne Kuxhausen Sign Name: DocuSigned by: Abrienne Kuxhausen Signer Name: Adrienne Kuxhausen Signing Reason: I approve this document Signing Time: 22-Nov-2019 15:28:45 EST 6E6B87C6B98740819F26B8D5A7D662CF | 22-Nov-2019 15:28:48 ES |
| BlackThorn<br>Therapeutics, Inc.<br>Representative | Print Name: Rezi Zawadzki Sign Name: | 22 - Nov. 2019 |





### **Document History**

| Version | Date | Author | Description |
|---|---|---|---|
| 0.1i | 08-Aug-2018 | Christopher Olson | Initial Draft |
| 0.2 | 16-Nov-2018 | Christopher Olson | Incorporated initial feedback, circulated for final review and finalization |
| 0.3 | 05-Mar-2019 | Christopher Olson | Incorporated feedback on shells and circulated for finalization |
| 1.0 | 10-Apr-2019 | Christopher Olson | Updated for finalization |
| 1.1 | 23-Sep-2019 | Christopher Olson | Added text for changes from planned analyses, as the planned PK analyses was not completed |



### **Table of Contents**

| Αŗ | provals | | 2 |
|----|----------|--------------------------------------------------|------|
| Do | cument | History | 3 |
| Ta | ble of C | Contents | 4 |
| 1. | Ov | rerview | 7 |
| 2. | Stı | ndy Objectives and Endpoints | 7 |
| | 2.1. | Study Objectives | 7 |
| | 2.1.1. | Safety Objectives | 7 |
| | 2.1.2. | Tolerability Objectives. | 7 |
| | 2.1.3. | Pharmacokinetic Objectives | 8 |
| | 2.1.4. | Efficacy Objectives | 8 |
| | 2.2. | Study Endpoints | 8 |
| | 2.2.1. | Primary Endpoint | 8 |
| | 2.2.2. | Secondary Endpoints | 8 |
| | 2.2.3. | Safety Endpoints | 8 |
| | 2.2.4. | Pharmacokinetic Endpoint | 8 |
| | 2.2.5. | Tolerability Endpoint | 9 |
| 3. | Ov | rerall Study Design and Plan | 9 |
| | 3.1. | Overall Design | 9 |
| | 3.2. | Sample Size and Power | 9 |
| | 3.3. | Study Population and Treatments Administered | 9 |
| | 3.4. | Method of Assigning Subjects to Treatment Groups | |
| | 3.5. | Blinding and Unblinding | . 10 |
| | 3.6. | Schedule of Events | . 10 |
| 4. | Sta | tistical Analysis and Reporting | . 12 |
| | 4.1. | Introduction | . 12 |
| | 4.2. | Interim Analysis and Data Monitoring | . 13 |
| 5. | An | alysis Populations | . 13 |
| | 5.1. | Statistical Definitions and Algorithms | . 13 |
| | 5.1.1. | Baseline | . 13 |
| | 5.1.2. | Adjustments for Covariates | . 13 |
| | 5.1.3. | Multiple Comparisons/Multiplicity | . 13 |
| | 5.1.4. | Handling of Dropouts or Missing Data | |
| | 5.1.5. | Analysis Visit Windows | |
| ΑD | -ST-33.0 | 4 Effective date: 30-Jun-2017 | |



| | 5.1.6. | Derived Variables | 14 |
|---|---|---|---|
| | 5.1.7. | Data Adjustments/Handling/Conventions | 14 |
| 6. | Stı | udy Subjects and Demographics | 16 |
| | 6.1. | Disposition of Subjects and Withdrawals | 16 |
| | 6.2. | Protocol Deviations | 16 |
| | 6.3. | Demographics and Other Baseline Characteristics | 16 |
| | 6.4. | Medical History | 16 |
| | 6.5. | Prior Medications | 17 |
| | 6.6. | Concomitant Medications | 17 |
| | 6.7. | Exposure and Study Drug Administration | 17 |
| 7. | Ef | ficacy Analysis | 17 |
| | 7.1. | Primary Efficacy Analysis | 17 |
| | 7.2. | Secondary Efficacy Analysis | 18 |
| 8. | Sa | fety and Tolerability Analysis | 18 |
| | 8.1. | Adverse Events | 18 |
| | 8.1.1. | Adverse Events Leading to Withdrawal | 19 |
| | 8.1.2. | Deaths and Serious Adverse Events | 19 |
| | 8.2. | Clinical Laboratory Evaluations | 19 |
| | 8.3. | Vital Signs | 19 |
| | 8.3.1. | Orthostatic Blood Pressure | 20 |
| | 8.4. | Electrocardiograms | 20 |
| | 8.5. | Pharmacokinetic Analysis | |
| | 8.6. | Columbia-Suicide Severity Rating Scale | 20 |
| | 8.7. | Impulsive Compulsive Disorders in Parkinson's Disease-Rating Scale | 20 |
| 9. | Ch | anges from Planned Analysis | 21 |
| 10. | Re | ferences | 22 |
| 11. | Ta | bles, Listings, and Figures | 22 |
| | 11.1. | Planned Table Descriptions | 24 |
| | 11.2. | Planned Figure Descriptions | 25 |
| | 11.3. | Planned Listing Descriptions | 26 |
| 12. | Ta | bles, Listings, and Figure Shells | 27 |
| | 12.1. | Standard Layout for all Tables, Listings, and Figures | |
| | 12.2. | Planned Table Shells | 28 |
| | 12.3. | Planned Figure Shells | 52 |





| 12.4. | Planned Listing Shells. | 53 |
|----------|------------------------------|----|
| Appendix | 1: Library of Abbreviations. | 78 |





### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for BlackThorn Therapeutics, Inc. protocol number NEP-PD-201 (*Phase 2a, Double-blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BTRX-246040 in Parkinson's Disease Subjects with Motor Fluctuations*), dated 31-Jul-2018. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents<sup>1, 2</sup>. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles for Clinical Trials<sup>3</sup>, International Conference on Harmonization; Statistical Principles for Clinical Trials: Addendum on Estimands and Sensitivity Analysis in Clinical Trials<sup>4</sup>. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association<sup>5</sup> and the Royal Statistical Society<sup>6</sup>, for statistical practice.

The planned analyses identified in this SAP will be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

The statistical plan described hereafter is an *a priori* plan. It will be submitted to file prior to any unblinded inferential or descriptive analysis of data pertaining to BlackThorn Therapeutics, Inc.'s study NEP-PD-201.

### 2. Study Objectives and Endpoints

### 2.1. Study Objectives

The purpose of this study is to assess the safety, tolerability, pharmacokinetics and efficacy of BTRX-246040 in subjects with Parkinson's Disease (PD) who have motor fluctuations and predictable early morning off periods.

### 2.1.1. Safety Objectives

• To evaluate the safety of single ascending doses of BTRX-246040 in PD subjects with motor fluctuations and predictable early morning off periods.

### 2.1.2. Tolerability Objectives

• To assess the tolerability of BTRX-246040 in PD subjects with motor fluctuations and predictable early morning off periods.



### 2.1.3. Pharmacokinetic Objectives

To evaluate the single-dose  $C_{max}$ ,  $T_{max}$ ,  $T_{10}$  and AUC of BTRX-246040.

To evaluate the relationship between clinical efficacy/response and plasma levels of

BTRX-246040 in PD subjects with motor fluctuations and predictable early morning off periods.

### 2.1.4. Efficacy Objectives

 To evaluate the effect of single ascending doses of BTRX-246040 on the clinical features of PD in levodopa-treated PD subjects with motor fluctuations and predictable early morning off periods.

### 2.2. Study Endpoints

### 2.2.1. Primary Endpoint

The primary endpoint of this study is the maximal change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III from pre-dose to post-dose on Day 1

### 2.2.2. Secondary Endpoints

The secondary endpoints of this study include the following:

- Duration of ON time on Day 1.
- Percentage of subjects that turn ON on Day 1.
- Time to ON on Day 1.
- Area under the curve for UPDRS Part III during the 8 hours of assessment on Day 1.
- Change from pre-dose dyskinesia rating (from the UPDRS Part III motor response and dyskinesia assessment).

### 2.2.3. Safety Endpoints

The safety endpoints of this study include the following:

- Adverse Events (AEs), AEs leading to discontinuation from the study drug, and serious AEs (SAEs).
- Change from baseline in clinical laboratory results, electrocardiogram (ECG) results, and vital signs.
- Neurological Exams.
- Columbia Suicide Severity Rating Scale (C-SSRS).

### 2.2.4. Pharmacokinetic Endpoint

• Pharmacokinetic profile will be evaluated by descriptive review of Cmax, Tmax, AUC, Elimination Half life parameters for BTRX-246040.



### 2.2.5. Tolerability Endpoint

Tolerability of BTRX-246040 will be assessed by the percentage of subjects who complete the protocol.

### 3. Overall Study Design and Plan

This is a phase 2a, double-blind, placebo-controlled study to investigate the safety, tolerability, pharmacokinetics, and efficacy of BTRX-246040 in PD subjects with motor fluctuations. A sample size of 8 subjects per cohort will be randomized to BTRX-246040 40 mg (1 capsule), 80 mg (2 capsules), 120 mg (3 capsules), or matching Placebo. Subjects must be between the ages of 30 and 76 and have a clinical diagnosis of PD with motor fluctuations and predictable early morning off periods.

The overall maximum study duration for an individual subject is expected to be approximately 36 days (including the 28 day screening period) with study drug treatment duration of 1 day. As per the schedule of events in <u>Table 2</u> subjects will be randomly assigned in a 6:2 ratio (BTRX-246040: Placebo) by cohort. After the 1 day treatment (including the 8 hour observation period), the study center will conduct a follow-up safety visit 7 days later (Day 8).

### 3.1. Overall Design

### 3.2. Sample Size and Power

No formal sample size calculations were calculated. A sample size of 8 subjects per group was deemed sufficient to evaluate the preliminary safety, tolerability, and efficacy of the different dose levels.

### 3.3. Study Population and Treatments Administered

The study will enroll approximately 24 subjects in a 6:2 ratio (BTRX-246040: Placebo) who have diagnosed PD with motor fluctuations and predictable early morning off periods. Additional subjects may be added to a cohort to better understand safety at a particular dose cohort.

This study involves a comparison of BTRX-246040 versus Placebo taken orally as a single dose in 3 sequential ascending dose cohorts. The planned dosing for each cohort is noted in Table 1.

**Table 1: Treatment Regimens** 

| Treatment Group | Regimen |
|---|---|
| BTRX-246040 | <ul> <li>Cohort 1 – 40 mg (1 capsule)</li> <li>Cohort 2 – 80 mg (2 capsules)</li> <li>Cohort 3 – 120 mg (3 capsules)</li> </ul> |
| Placebo | <ul> <li>Cohort 1 – (1 capsule)</li> <li>Cohort 2 – (2 capsules)</li> <li>Cohort 3 – (3 capsules)</li> </ul> |





| • |
|---|

Following completion of each cohort, unblinded safety, tolerability, efficacy and, if available, PK data will be reviewed by an unblinded Dosing Review Committee (DRC) to determine if it is safe to proceed to the next higher dose level.

### 3.4. Method of Assigning Subjects to Treatment Groups

In this parallel-group randomized phase 2a study, subjects who meet study entry criteria will be randomly assigned to receive BTRX-246040, or Placebo as described above at Visit 2. The randomization numbers will be assigned sequentially by cohort through a central interactive web-response system (IWRS) as subjects who meet eligibility criteria are enrolled into the study.

The randomization schedule will be prepared by Premier Research before the start of the study. No one involved in the clinical conduct will have access to the randomization schedule before official unblinding of treatment assignment. No subject will be randomized into the study more than once.

### 3.5. Blinding and Unblinding

BTRX-246040 and Placebo capsules and packaging will be identical to maintain the investigator, subject, and clinical study team member blinds.

All subjects, investigators, and study personnel involved in the conduct of the study, including data management, will be blinded to the treatment assignment with the exception of a prespecified independent statistician/programmer from Premier Research who will be involved in generation of the randomization code. The unblinded study personnel will not participate in study procedures or data analysis prior to unblinding of the study data which will be performed after database lock, but will be involved in preparing the unblinded report for the DRC.

Study personnel will endeavor to safeguard the integrity of the study blind to minimize bias in the conduct of the study. Treatment unblinding is discouraged but may be permitted in case of medical emergency only if that requires immediate knowledge of the subject's treatment assignment. The process of unblinding one subject should not jeopardize the validity and integrity of the whole study. If an Investigator, site personnel performing the assessments, or subject is unblinded, the subject must be discontinued from the study.

### 3.6. Schedule of Events

A detailed schedule of events for the study is provided in <u>Table 2</u>.

**Table 2: Schedule of Events** 

| SCRN | Treatment<br>Period | Follow-up or<br>Early<br>Termination | Unscheduled visits <sup>1</sup> |
|---|---|---|---|
| 1 | 2 | 3 | |
| -28 to 0 | 1 | 8 (±1) | |
| X | | | |
| X | | | |
| X | | | |
| X | X | X | X |
| X | X | X | X |
| X | | X | X |
| X | | X | |
| X | X | X | X |
| X | | | |
| | X | X | X |
| X | | | |
| X | | | |
| X | | | |
| | X | X | X |
| X <sup>4</sup> | X <sup>5</sup> | | |
| X <sup>4</sup> | X <sup>5</sup> | | |
| X | | | |
| X | X | X | X |
| X | | | |
| | 1 -28 to 0 X X X X X X X X X X X X X X X X X X X | SCRN Period 1 | SCRN Treatment Period Early Termination 1 2 3 -28 to 0 1 8 (±1) X X X X X |

<sup>&</sup>lt;sup>1</sup> Unscheduled visits may be conducted at any time for safety reasons and/or for any other reason.

<sup>&</sup>lt;sup>2</sup> Vital signs include supine (at least 5 min) and standing (after approximately 2 min) BP and pulse rate, body temperature and body weight. At Day 1, 3 sets each of supine and standing BP and pulse rate will be measured at least 15-20 minutes apart at pre-dose and will be measured once at 2, 4, 6, and 8 hours after dosing.

<sup>&</sup>lt;sup>3</sup> Height will be measured only once, at Screening. Body weight will be measured once per visit.

<sup>&</sup>lt;sup>4</sup> At screening, UPDRS Part III and dyskinesia rating should be done in the OFF and the ON state. This can be done in either the practically defined OFF state or after a subject wears OFF following a levodopa dose.

<sup>&</sup>lt;sup>5</sup> At Day 1, UPDRS Part III and dyskinesia rating will be conducted in the OFF state Pre-dose and every 30 minutes for 4 hours and then hourly for another 4 hours (or until subject turns OFF) following study drug administration. If the subject remains ON after 8 hours, they should be called the next morning to record the time they turned OFF, and the time they took their first regularly scheduled anti-parkinsonian medications after study drug, to a maximum of 24 hours



| Laboratory Evaluation | X | | X | X |
|-------------------------------------------------------|---|---|---|---|
| Urine drug screen | X | | | |
| Approval via Enrollment Authorization Committee (EAC) | X | | | |
| Randomization | | X | | |
| Study Drug administered | | X | | |
| Adverse Events | | X | X | X |
| BTRX-246040 pharmacokinetics <sup>6</sup> | | X | | |
| Time to ON and duration of ON recorded | | X | | |
| Drug accountability | | X | | |

BTRX-246040 pharmacokinetics to be collected pre-dose and 30, 60, 120, 240, and 480 minutes after study drug

### 4. Statistical Analysis and Reporting

All final, planned analyses identified in this SAP will be performed after the study database has been locked and treatment codes have been unblinded.

### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed using SAS® (release 9.4 or higher. If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous variable summaries will include the number of subjects (n) with non-missing values, mean, standard deviation (SD), median, minimum, and maximum.

Categorical variable summaries will include the frequency and percentage of subjects that are in the particular category or each possible value. In general the denominator for the percentage calculation will be based upon the study population for the specified treatment group and overall, unless otherwise specified. The denominator for by-visit displays will be the number of subjects in the relevant study population and treatment with non-missing data at each visit.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data and measures of spread (SD) will be reported to 2 degrees of precision more than the observed data. Percentages will be presented to 1 decimal place, unless otherwise specified.





### 4.2. **Interim Analysis and Data Monitoring**

No interim analysis is currently planned. If an interim analysis is planned in the future, this will be amended in protocol and in the SAP text as applicable. Safety of planned cohorts will be evaluated by the DRC per section 9.7 of the protocol.

### 5. **Analysis Populations**

The following 2 analysis populations are planned for this study:

- Modified Intent-to-Treat Population (mITT): Includes all randomized subjects who received at least one dose of study drug and have at least 1 post-baseline scoring of motor activity. In accordance with the intent-to-treat principle, all subjects will be kept in their randomized treatment group. The mITT population will serve as the primary population for efficacy evaluations.
- Safety Analysis Population (SAF): Includes all subjects who have received study drug. All subjects will be evaluated according to actual treatment received. The safety population will serve as the primary population for safety evaluations.

Inclusion in the analysis populations described above will be determined prior to database lock.

### 5.1. **Statistical Definitions and Algorithms**

### 5.1.1. Baseline

The last non-missing observation recorded on or before the first dose of study drug will be used as the baseline observation for all calculations of change from baseline.

### 5.1.2. Adjustments for Covariates

No planned covariates will be included in any planned analyses. Exploration of additional covariates will be considered as data becomes available post database lock.

### 5.1.3. Multiple Comparisons/Multiplicity

There will be no adjustments for multiple comparisons for efficacy or safety endpoints.

### 5.1.4. Handling of Dropouts or Missing Data

There will be no imputation for efficacy or safety endpoints.





### **5.1.5.** Analysis Visit Windows

In general, analysis of all variables for this study will use the nominal visit or time point as collected in the eCRF/database. Scheduled visits will be selected over unscheduled visits. Unscheduled visits will be presented in data listings.

### 5.1.6. Derived Variables

- Study Day = Assessment Date Date of First Dose + 1
- Change from Baseline = Value Post-Baseline Value at Baseline
- % Change from Baseline = 100 \* Change from Baseline / Value at Baseline
- Duration of ON time on Day 1 = First returned to OFF state Datetime (UPDRS2) or DFUP CRF Page) - First reported ON state Datetime (UPDRS2 CRF Page)
- Time to ON on Day 1 = First reported ON state Datetime (UPDRS2 CRF Page) -Study drug administration Datetime (EX1 CRF Page)
- UPDRS Part III Score = Summation of all items in motor examination (14-item rating scale), each item scored from 0 (Normal) to 4 (Most severe). If any item is missing, the total score will be missing.
- Adverse events beginning with the initial dose of IP or during subsequent duration of their enrollment in the study will be considered treatment-emergent AEs (TEAEs)

It is expected additional derived variables will be needed, but the SAP will not be amended unless they are part of the primary or secondary endpoints in the study.

### 5.1.7. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

In general for quantitative laboratory values reported as '<' or '\(\section\), the lower limit of quantitation (LLOQ) or limit of detection (LOD), one-half of the reported value (i.e., LLOQ, LOD) will be used for analysis. For quantitative laboratory values reported as '>' or  $\geq$ , the upper limit of quantitation (ULOQ), the reported value (i.e., ULOQ) will be used for analysis.





For analysis purposes, repeat laboratory test results will not be used unless the original laboratory value is missing or indicated as invalid, in which case the first non-missing repeat laboratory value will be used for data analysis.

Adverse events and Medical History will be coded using the MedDRA thesaurus. Concomitant and Prior medications will be coded using WHO Drug Dictionary (WHO-DD).

If partial dates occur for AEs or medications, the convention for replacing missing dates for analyses is as follows:

### For partial start dates:

- If the year is unknown, then do not impute the date but assign a missing value.
- If the month is unknown, then:
  - o If the year matches the year of the randomization date, then impute the month and day of the randomization date.
  - o Otherwise, assign 01 January
- If the day is unknown, then:
  - o If the month and year match the month and year of the randomization date, then impute the day of the first study drug administration date.
  - Otherwise, assign 01.

### For partial end dates:

- If the year is unknown, then do not impute the date but assign a missing value.
- If the month is unknown, then assign the last day of the year 31 December.
- If the day is unknown, then assign the last day of the month.

After implementing the rules above, to determine whether AEs (or medications) with missing start or stop dates are pretreatment or on/after treatment, the following strategy will be used:

- 1. If the start date and stop date are both missing, then the most conservative approach is taken and the AE (or medication) is considered to be treatment emergent (or concomitant).
- 2. If the start date is missing but the stop date is not missing and is after the day of study drug administration, then the most conservative approach is taken and the AE (or medication) is considered to be treatment emergent (or concomitant).
- 3. If the start date is missing but the stop date is not missing and is on or before the day of study drug administration, then the AE (or medication) is considered to be





before treatment (or prior).

If the start date is not missing but the stop date is missing, then the most conservative approach is taken. Medication is considered to be concomitant and AEs are considered to be treatment-emergent.

A treatment related AE is any AE with a relationship to the study drug of "Possibly Related", "Probably Related" or "Related". Any AE with a missing relationship will be analyzed as treatment related. If an AE has a missing severity, it will be imputed as "Severe".

### **Study Subjects and Demographics** 6.

### 6.1. **Disposition of Subjects and Withdrawals**

Disposition will include tabulations by treatment group and overall of the number of subjects randomized into each treatment group, the number of subjects who received treatment, tabulated reasons for discontinuation from the study, and number of subjects in each analysis population.

A by-subject listing of all disposition information will be presented.

### 6.2. **Protocol Deviations**

A by-subject listing of all protocol deviations and their category, description and type will be presented.

### 6.3. **Demographics and Other Baseline Characteristics**

Descriptive summaries of demographic (age, gender, race, ethnicity) and other baseline characteristics (height, weight and BMI) will be provided for all subjects by treatment group and overall. These tabulations will be repeated for mITT and SAF populations. Any physical examination/neurological exam findings will be recorded as medical history or AEs and will be summarized as specified in Section 6.4 or 8.1.

All demographic and other baseline characteristics will be presented in subject listings.

### 6.4. **Medical History**

Subjects reporting various medical histories, grouped by MedDRA system organ class (SOC) and preferred term (PT) will be tabulated for the SAF population.

A by-subject listing of all medical and PD history will be presented.





### 6.5. Prior Medications

Subjects taking prior medications, coded using WHO-DD Enhanced Version Sep. 2017 will be tabulated by Anatomical Therapeutic Chemical (ATC) classification level 4 and preferred term. A prior medication is any non-protocol specified drug or substance administered prior to first date of study drug whether or not it was stopped before administration.

A by-subject listing of all prior and concomitant medications will be presented.

### 6.6. Concomitant Medications

Concomitant medications will be tabulated similarly to Prior medications. A concomitant medication is any non-protocol specified drug or substance administered during participation in the study on or after first date of study drug. A medication can be considered both concomitant and prior if the subject took medication prior to the study and continued taking it after first study drug administration.

### 6.7. Exposure and Study Drug Administration

A by subject listing will be provided for all drug exposure and study drug administration information collected.

### 7. Efficacy Analysis

All efficacy variables will be summarized using the mITT population as the primary population of interest, unless otherwise specified.

### 7.1. Primary Efficacy Analysis

The primary efficacy endpoint of this study is the maximal change in UPDRS Part III Total Score from pre-dose to post-dose on Day 1 (collected every 30 minutes for 4 hrs, then hourly for 4 more hours) in all subjects. The mean maximal change will be presented along with its standard deviation, by treatment group. Data for all BTRX-246040 subjects pooled across cohorts will be compared with data for all Placebo subjects pooled across cohorts.

The observed value and change from baseline will be summarized descriptively for UPDRS Part III Total Score at each Day 1 time point, in addition to the maximal change described above. A scatter plot of the maximal change in UPDRS Part III Total Score will also be presented.





### 7.2. **Secondary Efficacy Analysis**

The secondary endpoints consist of the following:

- Duration of ON time on Day 1
- Percentage of subjects that turn ON on Day 1
- Time to ON on Day 1
- AUC for UPDRS Part III during the 8 hours of assessment on Day 1
- Change from pre-dose dyskinesia rating (from the UPDRS Part III motor response and dyskinesia assessment)

For continuous results noted above, the observed value and change from baseline for each time point will be summarized by treatment group. For categorical results, the frequency and percentage of subjects will be provided. Graphical displays for these endpoints will be created as applicable, including a scatter plot of UPDRS by time point and treatment.

### 8. Safety and Tolerability Analysis

Safety will be evaluated from reported TEAEs, changes in clinical laboratory values, changes in vital signs, ECG, physical examination results, neurological examination, and the C-SSRS. No formal inferential analyses will be conducted for safety outcomes, unless otherwise noted. Unless otherwise specified, all safety analyses will be conducted on the SAF population.

### 8.1. **Adverse Events**

All AEs and SAEs will be coded using the MedDRA v20.1 thesaurus. Adverse event analyses will include TEAEs, defined as AEs which start after the first dose of study medication. The frequency and percentage of subjects reporting TEAEs, grouped by MedDRA SOC and PT, will be tabulated by treatment group for the SAF. Such summaries will be displayed for the following:

- TEAEs by SOC and PT
- TEAEs by SOC, PT, and severity
- TEAEs by SOC, PT, and relationship to the study medication
- TEAEs leading to death by SOC, and PT
- SAE TEAEs other than deaths by SOC, and PT
- AEs leading to premature discontinuation by SOC, and PT
- Listing of non-TEAEs

In the case of multiple occurrences of the same AE within the same subject, each subject will only be counted once for each preferred term. In the summaries showing severity and relationship to study medication the event with the maximum severity or strongest





relationship will be reported. If a particular event is missing the severity and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = related).

Missing and partially missing AE start and/or stop dates will be imputed for the purpose of statistical analysis, according to the specifications described in Section 5.1.7.

In the AE data listings, all AEs will be displayed and TEAEs will be flagged. In the event the number of TEAEs is low from the tabulations above, only listings will be provided.

### 8.1.1. Adverse Events Leading to Withdrawal

A summary of incidence rates (frequencies and percentages) of AEs leading to withdrawal of study drug, by treatment group, SOC, and preferred term will be prepared.

### 8.1.2. Deaths and Serious Adverse Events

Any deaths that occur during the study will be listed.

Serious adverse events will be listed and also tabulated by system organ class and preferred term and presented by treatment.

### 8.2. Clinical Laboratory Evaluations

Descriptive summaries of actual (absolute) values and changes from baseline will be presented for each clinical laboratory analyte by treatment group.

The number of subjects with clinical laboratory values below, within, or above the normal range by time point will be tabulated for each clinical laboratory analyte by treatment group. These shift tables will tabulate the number and proportion of subjects from baseline to post-baseline categories of low, normal or high.

By-subject listings of laboratory analytes will be presented. Any out-of-range values that are identified by the investigator as being clinically significant will be shown on this listing.

Pregnancy and urine drug screen test results will be listed.

### 8.3. Vital Signs

Descriptive summaries of actual values and changes from baseline will be calculated for systolic blood pressure, diastolic blood pressure, pulse, respiratory rate, BMI, body weight, and oral body temperature. This summary will be presented by treatment group. Height and Weight at screening will be used to calculate BMI.

A by-subject listing of all vital sign measurements will be presented.





### 8.3.1. Orthostatic Blood Pressure

A separate summary with descriptive statistics of orthostatic blood pressure and pulse will be presented by time point, including values and change from baseline. The average of the three orthostatic BP and pulse measurements will be used for comparison to all post-treatment measurements to minimize the impact of biological variability and to serve as a more reliable baseline.

Additionally, the number and percentage of subjects with abnormal drops will also be shown. A drop in systolic blood pressure of > 20 mmHg, or in diastolic blood pressure of  $\geq$  10 mmHg upon standing will be considered abnormal.

A by-subject listing of orthostatic blood pressures will be presented.

### 8.4. **Electrocardiograms**

Descriptive summaries will be presented for ECG measures of PR interval, QRS interval, OT interval, OTc interval (both correction methods), RR interval and HR. These summaries will be presented by treatment group at each visit.

The frequency and percentage of subjects with normal and abnormal ECG results will be summarized by treatment group at each visit. A by-subject listing of all ECG measures and incidences of abnormalities will be presented.

### 8.5. Pharmacokinetic Analysis

Individual concentration vs actual time data will be used to estimate the PK parameters (Cmax, Tmax, T1/2, AUC) of BTRX-246040 by standard non-compartmental methods for each subject in the SAF population.

For PK data, all values below the limit of quantification (BLQ) will be set to 0 for summary statistics and graphs. Individual concentrations of BTRX-256040 will be summarized at each time point using descriptive statistics. Individual concentration plots and mean data graphs will be produced. All graphs will be presented using both linear and semi-logarithmic scales.

All BTRX-256040 concentration data will be presented in a by-subject listing.

### 8.6. **Columbia-Suicide Severity Rating Scale**

All measures of suicidal ideation and behavior collected on the C-SSRS will be listed by subject.

### 8.7. Impulsive Compulsive Disorders in Parkinson's Disease-Rating Scale

The frequency and percentage of subjects with positive response ("rarely" or higher) for





each disorder will be tabulated by treatment group and visit. Additionally, the total Impulsive Control Disorder score and total QUIP-RS score will also be presented with descriptive statistics by treatment group and visit (both actual values and changes from baseline). All scales will be presented in a by-subject listing with the individual questions and total scores shown.

### 9. Changes from Planned Analysis

- The relationship between clinical efficacy/response and plasma levels of BTRX-246040 in PD subjects with motor fluctuations and predictable early morning off periods was not analyzed.
- The planned PK analyses of Cmax, Tmax, T1/2, AUC were not calculated.

There are no additional changes to the planned analyses specified in the protocol.



### 10. References

- 1. BlackThorn Therapeutics, Inc. protocol number NEP-PD-201, *Phase 2a, Double-blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BTRX-246040 in Parkinson's Disease Subjects with Motor Fluctuations*, dated 31-Jul-2018
- 2. BlackThorn Therapeutics, Inc. eCRF NEP-PD-201, dated 21-Sep-2018, v1.0
- 3. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 4. US Federal Register. (2017) International Conference on Harmonization; Statistical Principles for Clinical Trials: Addendum on Estimands and Sensitivity Analysis in Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. FDA-2017-D-6113-0002]. October 31, 2017.
- 5. ASA. (2018) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 14, 2018. http://www.amstat.org/about/ethicalguidelines.cfm
- 6. RSS. (2014) The Royal Statistical Society: Code of Conduct, June 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf..

### 11. Tables, Listings, and Figures

All listings, tables, and graphs will have a header showing the sponsor's company name and protocol, the footer indicates the file name, path, and the source of the data (listing number).

### **General Reporting Conventions:**

- All tables and data listings will be developed in landscape orientation.
- Specialized text styles, such as bolding, italics, borders, shading, superscripted
  and subscripted text will not be used in tables and data listings unless they add
  significant value to the table, figure, or data listing.
- Only standard keyboard characters should be used in tables and data listings. Special characters, such as nonprintable control characters, printer-specific characters, or font specific characters, will not be used on a table, figure, or data listing. Hexadecimal character representations are allowed (e.g., μ, α, β).
- All titles will be centered on a page. The ICH numbering convention is to be used for all outputs.
- All footnotes will be left justified and at the bottom of a page.
- Missing values for both numeric and character variables will be presented as



blanks in a table or data listing. A value of zero may be used if appropriate to identify when the frequency of a variable is not observed.

- All date values will be presented as ddmmmyyyy (e.g., 29AUG2011) format. A 4-digit year is preferred for all dates.
- If applicable, all observed time values will be presented by using a 24-hour clock HH:MM:SS format (e.g., 01:35:45 or 11:26). Seconds should only be reported if they were measured as part of the study.
- All tables and data listings will have the name of the program, the location, and a run date and time stamp on the bottom of each output.

### **Population Summary Conventions**

- Population sizes may be presented for each classification factor as totals in the column header as (N=xxxx), where appropriate.
- Population sizes shown with summary statistics are the sample size (n) of subjects with non-missing values.
- All population summaries for categorical variables will include all categories that were planned and for which the subjects may have had a response. Percentages corresponding to null categories (cells) will be suppressed, however counts and percentages of missing values may be needed.
- All population summaries for continuous variables will include: N, mean, median, SD, minimum, and maximum. Other summaries (e.g., number missing) may be used as appropriate.
- All percentages are rounded and reported to a single decimal point (xx.x %). A percentage of 100% will be reported as 100%. No value of 0% will be reported. Any computation of percent that results in 0% is to be presented as a 0.





### 11.1. Planned Table Descriptions

The following are planned summary tables for protocol number NEP-PD-201. The table numbers and page numbers are place holders only and will be determined when the tables are produced.

| Table Number | Population | Table Title |
|---|---|---|
| | s and Baseline Tables | |
| 14.1.1 | SCREEN | Study Populations and Subject Disposition |
| 14.1.2.1 | SAF | Demographics |
| 14.1.2.2 | mITT | Demographics Demographics |
| 14.1.3 | SAF | Medical History |
| 14.1.4 | SAF | Concomitant Medications |
| 14.1.5 | SAF | Prior Medications |
| 14.2 Efficacy and | | THO MEDICALIONS |
| 1 1.2 Efficacy and 1 | Tubles | Summary of UPDRS Part III Total Score pre-dose to post- |
| 14.2.1.1 | mITT | dose on Day 1 |
| 14.2.1.2 | mITT | AUC of UPDRS Part III Total Score |
| 14.2.2 | mITT | Summary of Dyskinesia Rating on Day 1 |
| 14.2.3 | mITT | Summary of Duration of ON and Time to ON on Day 1 |
| 14.2.4 | mITT | Summary of Pharmacokinetic Parameters |
| 14.3 Safety and To | | |
| 14.3.1 Displays of | | |
| 14.3.1.1 | SAF | Summary of all TEAEs |
| 14.3.1.2 | SAF | TEAEs by SOC and Preferred Term |
| 14.3.1.3 | SAF | TEAEs by SOC, Preferred Term and Severity |
| | | TEAEs by SOC, Preferred Term and Relationship to Study |
| 14.3.1.4 | SAF | Medication |
| - | | TEAEs leading to discontinuation by SOC and Preferred |
| 14.3.1.5 | SAF | Term |
| 14.3.1.6 | SAF | TESAEs other than deaths by SOC and Preferred Term |
| 14.3.1.7 | SAF | TEAEs leading to death by SOC and Preferred Term |
| 14.3.2 Laboratory | Safety Data | • |
| 14.3.2.1 | SAF | Summary of Clinical Chemistry by Study Visit |
| 14.3.2.2 | SAF | Summary of Hematology by Study Visit |
| 14.3.2.3 | SAF | Summary of Urinalysis by Study Visit |
| 14.2.2.4 | SAF | Summary of Coagulation by Study Visit |
| 14.3.2.5 | SAF | Shifts from Baseline of Clinical Chemistry by Study Visit |
| 14.3.2.6 | SAF | Shifts from Baseline of Hematology by Study Visit |
| 14.3.2.7 | SAF | Shifts from Baseline of Urinalysis by Study Visit |
| 14.3.2.8 | SAF | Shifts from Baseline of Coagulation by Study Visit |
| 14.3.3 Vital Signs | and ECG Data | <u> </u> |
| 14.3.3.1 | SAF | Summary of Vital Signs by Study Visit |
| | | Summary of Orthostatic Blood Pressure and Pulse by |
| 14.3.3.2 | SAF | Study Visit |
| | | Incidence of Abnormal Orthostatic Blood Pressure by |
| 14.3.3.3 | SAF | Study Visit |
| 14.3.3.4 | SAF | Summary of ECG Parameters by Study Visit |
| 14.3.3.5 | SAF | Incidence of Abnormal ECG by Study Visit |
| 14.3.4 Other Safet | y Data | |
| 14.3.4.1 | SAF | Summary of Impulsive Control Disorder and QUIP-RS by |
| | • | |



| Study Visit |
|-------------|
| Study Visit |

### 11.2. Planned Figure Descriptions

The following are planned summary figures for protocol number NEP-PD-201. The figure numbers and page numbers are place holders only and will be determined when the figures are produced.

| Figure Number | Population | Figure Title |
|---|---|---|
| 14.2 Efficacy Figur | res | |
| 14.2.1 | mITT | AUC of UPDRS Part III Total Score |
| | | Scatter Plot of maximal change in UPDRS Part III Total |
| 14.2.2 | mITT | Score |
| 14.2.3 | mITT | Scatter Plot of UPDRS Part III Total Score by timepoint |
| 14.3 Safety Figure | S . | |
| 14.3.1 | SAF | Scatter Plot of serum concentration linear |
| 14.3.2 | SAF | Scatter Plot of serum concentration (logarithmic) |





### 11.3. Planned Listing Descriptions

The following are planned data and subject data listings for protocol number NEP-PD-201.

| T' 4' NL 1 | D1 4' | T' ' T'' |
|---|---|---|
| Listing Number | Population | Listing Title |
| 16.2.1 Subject Dispo | | A ' 44 A 1-' D -14' 1T 4 4 A |
| 16.2.1.1 | SCREEN | Assignment to Analysis Populations and Treatment Arm |
| 16.2.1.2 | SCREEN | Study Completion Status and Reasons for Discontinuation |
| 16.2.1.3 | SCREEN | Inclusion and Exclusion Criteria |
| 16.2.2 Protocol Devi | | |
| 16.2.2.1 | mITT | Protocol Deviations |
| | s and Other Baseline C | |
| 16.2.4.1 | SAF | Demographics |
| 16.2.4.2 | SAF | Medical and PD History |
| 16.2.4.3 | SAF | Concomitant and Prior Medications |
| | re and Concentration D | |
| 16.2.5.1.1 | SAF | Drug Accountability |
| 16.2.5.1.2 | SAF | Study Drug Administration |
| 16.2.5.2 | SAF | Serum Concentration of BTRX-246040 |
| 16.2.6 Efficacy Listi | | |
| 16.2.6.1 | mITT | Unified Parkinson's Disease Rating Scale (Part III) |
| 16.2.6.2 | mITT | Total UPDRS Score (Part III) and Dyskinesia Rating |
| 16.2.6.3 | mITT | Time to and Duration of ON state |
| 16.2.7 Adverse Even | nt Listings | |
| 16.2.7.1 | SAF | Treatment-Emergent Adverse Events |
| 16.2.7.2 | SAF | Serious Adverse Events |
| 16.2.7.3 | SAF | Adverse Events Leading to Discontinuation |
| 16.2.7.4 | SAF | Listing of Deaths |
| 16.2.8 Laboratory D | oata Listings | |
| 16.2.8.1 | SAF | Clinical Chemistry |
| 16.2.8.2 | SAF | Hematology |
| 16.2.8.3 | SAF | Urinalysis |
| 16.2.8.4 | SAF | Coagulation |
| 16.2.8.5 | SAF | Urine Drug Screen |
| | l Observations and Me | |
| 16.2.9.1 | SAF | Vital Signs |
| 16.2.9.2 | SAF | Electrocardiogram |
| 16.2.9.3 | SAF | Physical Examination |
| 16.2.9.4 | SAF | Neurological Examination |
| 16.2.9.5 | SAF | Columbia-Suicide Severity Rating Scale (C-SSRS) |
| | | Questionnaire for Impulsive-Compulsive Disorders in |
| 16.2.9.6 | SAF | Parkinson's disease Rating Scale (QUIP-RS) |
| 16.2.9.7 | SAF | Montreal Cognitive Assessment (MoCA) |
| 16.2.9.8 | SAF | Beck Depression Inventory-II |
| 16.2.9.9 | SAF | Modified Hoehn and Yahr scale |
| 10.2.7.7 | ~111 | 1.15 dilled 110 dilli dild 1 dill 50 die |

Statistical Analysis Plan, Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311



## 12. Tables, Listings, and Figure Shells

# 12.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all Tables, Listings, and Figures in support of this study. Note that programming notes may be added if appropriate after each TLF shell as noted by {}.

### Standardized Layout

| BlackThorn Therapeutics, Inc.<br>Protocol NEP-PD-201 | Page xx of xx |
|---|---|
| <table, figure="" listing,=""> xx.x.x<br/><title figure="" listing="" of="" or="" table="">&lt;br&gt;&lt;Study Population and if applicable subgroup Description&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Body of Table, Listing or Figure&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Note: &lt;&lt;i&gt;Note&lt;/i&gt;: If directly Applicable&gt; Footnote 1 &lt;if applicable&gt; Footnote 2 &lt;if applicable&gt; Footnote n &lt;if applicable&gt; Footnote n &lt;if applicable&gt; Source: Listings xx.x.x, xx.x.x &lt;if applicable&gt; T:\BlackThorn\NEP-PD-201\\xxxxxx.ss run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;/tbody&gt;&lt;/table&gt;</title></table,> | |



## 12.2. Planned Table Shells

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Table 14.1.1 Study Populations and Subject Disposition All Screened Subjects

 FINAL

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| Status or | 40 mg | 80 mg | 120 mg | Placebo |
| Variable/Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Screened for Eligibility | × | × | × | × |
| Randomized | ×× | X | X | × |
| mITT Population [1] | × | × | × | × |
| SAF Population [2] | × | × | × | × |
| Completed Study Treatment | (%X:X%) | (%x.xx) xx | xx (xx.x%) | (%x.x%) xx |
| Early Discontinuation | (%x.x%) | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx |
| Reason for Early Discontinuation [3] | | | | |
| Physician decision | (%x.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawal by subject | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Study terminated by sponsor | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse event | (%x.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost to follow-up | (%x.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | (%x.xx) xx | (%x.x%) | (%x.xx) xx |

Note: Percentages are based on the number of subjects in the SAF Population. Assigned/planned treatment groups are presented.

[1] The Modified Intent-to-Treat Population (mITT) includes all randomized subjects who received at least one dose of study drug and have at least 1 post-baseline scoring of motor activity. All subjects will be evaluated according to assigned treatment.

[2] The Safety Population (SAF) includes all subjects who have received study drug. All subjects will be evaluated according to actual treatment type received.

[3] Percentages are based off of number of early terminations per applicable treatment column.

{Programming Note: If treatment/bottle mix-up occurs and subject takes one or more incorrect pills, please footnote this in this table with surrounding details} SOURCE: Listings xx.x.x, xx.x.x

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY



BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Safety Population Demographics Table 14.1.2.1

FINAL 

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| Variable | 40 mg | 80 mg | 120 mg | Placebo |
| Statistics or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Age (years) | | | | |
| :<br>:<br>: | × | × | × | × |
| Mean | xx.x | xx.x | XX.X | XX.X |
| Standard Deviation | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | xx.x | xx.x | xx.x |
| Minimum, Maximum | xx, xx | xx, xx | xx, xx | xx, xx |
| Gender | | | | |
| Male | (%x:x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Female | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx |
| Race | | | | |
| American Indian or Alaska Native | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Asian | x (xx.x%) | xx (xx.x%) | (%x.x%) xx | xx (xx.x%) |
| Black or African American | (%x.xx) xx | xx (xx.x%) | (%x.x%) xx | xx (xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| White | x (xx.x%) | xx (xx.x%) | (%x.x%) xx | xx (xx.x%) |
| More than one race | (%X.XX) XX | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received.

SOURCE: Listings xx.x.x, xx.x.x T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMIMMYYYY at HH:MM on data extracted on DDMIMMYYYY





 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Demographics Safety Population Table 14.1.2.1

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| Variable | 40 mg | 80 mg | 120 mg | Placebo |
| Statistics or Category | (xx=N) | (N=xx) | (N=xx) | (N=xx) |
| Ethnicity | | | | |
| Hispanic or Latino | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Hispanic or Latino | (%x.x%) | xx (xx.x%) | xx (xx.x%) | (%x.x%) xx |
| Height (cm) | | | | |
| L | × | × | ×× | X |
| Mean | XXX.X | XXX.X | xxx.x | XXX.X |
| Standard Deviation | XXX.XX | xx.xx | XXX.XX | XXX.XX |
| Median | XXXX.X | xxx.x | xxx.x | XXX.X |
| Minimum, Maximum | xxx, xxx | xxx, xxx | xxx, xxx | xxx, xxx |
| Weight (kg) | | | | |
| L | × | ×× | ×× | X |
| Mean | XXX.XX | xxx.xx | XXX.XX | XXX.XX |
| Standard Deviation | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| Median | XXX.XX | xxx.xx | XXX.XX | XXX.XX |
| Minimum, Maximum | XXX.X, XXX.X | xxx.x, xxx.x | xxx.x, xxx.x | XXX.X, XXX.X |

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. SOURCE: Listings xx.x, xx.x, xx.x.x T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY





FINAL 

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Demographics Safety Population Table 14.1.2.1

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| Variable | 40 mg | 80 mg | 120 mg | Placebo |
| Statistics or Category | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| BMI (kg/m2) | × | × | ×× | × |
| u | XX.XXX | XX.XXX | XX.XXX | xx.xxx |
| Mean | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Standard Deviation | xx.xx | XX.XXX | XX.XXX | xx.xxx |
| Median | XX.XX, XX.XX | xx.xx, xx.xx | xx.xx, xx.xx | XX.XX, XX.XX |
| Minimum, Maximum | | | | |
| Years of education (yrs) | | | | |
| L | ×× | × | × | × |
| Mean | xxx.x | xxx.x | xxx.x | xxx.x |
| Standard Deviation | xx.xx | xx.xx | xxx.xx | xxx.xx |
| Median | xxx.x | xxx.x | xxx.x | xxx.x |
| Minimum, Maximum | xxx, xxx | xxx, xxx | xxx, xxx | xxx, xxx |

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received.

SOURCE: Listings xx.x.x, xx.x.x

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY

Table 14.1.2.2

Demographics Modified Intent-to-Treat Population

(Programming Note: Repeat 14.1.2.1 with mITT population, update footnote to indicate planned treatment groups are presented)





FINAL 

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Safety Population **Medical History** Table 14.1.3

| System Organ Class [1] | BTRX-246040<br>40 mg<br>(N=xx) | BTRX-246040<br>80 mg<br>(N=xx) | BTRX-246040<br>120 mg<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Number of subjects with at least one medical history | (XX.X%) | (XX.XX) | (%x.x%) xx | (%x:x%) xx |
| SOC 1 | (%x:x%) | xx (xx.x%) | (%x.xx) xx | (%x:xx) xx |
| PT1 | xx (xx.x%) | xx (xx.x%) | (%x:x%) xx | xx (xx.x%) |
| PT 2 | xx (xx.x%) | x (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 3 | xx (xx.x%) | xx (xx.x%) | (%x.x%) xx | xx (xx.x%) |
| SOC 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 1 | xx (xx.x%) | xx (xx.x%) | (%x:x%) | xx (xx.x%) |
| PT 2 | (%x.xx) xx | xx (xx.x%) | (%x.x%) xx | (%x.xx) xx |

{Repeated for all applicable SOC/PT combinations}

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. Subjects were counted only once for each System Organ Class and Preferred Term. [1] Medical History was coded using MedDRA version 20.1.

SOURCE: Listings xx.x.x, xx.x.x

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY





FINAL 

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Table 14.1.4

Concomitant Medications Safety Population

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | | i |
|---|---|---|---|---|---|
| ATC [1] | 40 mg | 80 mg | 120 mg | Placebo | |
| Preferred Term | (N=xx) | (x=n) | (N=xx) | (N=xx) | ı |
| Number of subjects with at least one concomitant medication | xx (xx.x%) | xx (xx.x%) | (%x.x%) | (xx.x%) | |
| ATC 1 | xx (xx.x%) | xx (xx.x%) | (%x:x%) xx | xx (xx.x%) | |
| Medication 1 | xx (xx.x%) | (%x.x%) xx | xx (xx.x%) | xx (xx.x%) | |
| Medication 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | xx (xx.x%) | (%x.x%) | xx (xx.x%) | xx (xx.x%) | |
| ATC 2 | | | | | |
| Medication 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Medication 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | xx (xx.x%) | x (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

{Repeated for all applicable ATC/PT combinations}

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. Subjects were counted only once for each Anatomical Therapeutic Chemical (ATC) or Preferred Term. A concomitant medication is any non-protocol specified drug or substance administered during participation in the study on or after first date of study

[1] Medications were coded using WHO-DD (Enhanced version Sep. 2017), ATC Level 4

SOURCE: Listings xx.x.x, xx.x.x

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY

Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311 Statistical Analysis Plan,



 FINAL

BlackThorn Therapeutics, Inc.

Protocol NEP-PD-201

**Prior Medications** Safety Population **Table 14.1.5** 

| ATC [1]<br>Preferred Term | BTRX-246040<br>40 mg<br>(N=xx) | BTRX-246040<br>80 mg<br>(N=xx) | BTRX-246040<br>120 mg<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Number of subjects with at least one prior medication | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| Medication 1 | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) |
| Medication 2 | xx (xx.x%) | (%x:xx) xx | xx (xx.x%) | (%x.xx) xx |
| | xx (xx.x%) | (%x.x%) xx | xx (xx.x%) | xx (xx.x%) |
| ATC 2 | | | | |
| Medication 1 | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx |
| Medication 2 | xx (xx.x%) | (%x:x%) xx | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

{Repeated for all applicable ATC/PT combinations}

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. Subjects were counted only once for each Anatomical Therapeutic Chemical (ATC) or Preferred Term. A prior medication is any non-protocol specified drug or substance administered prior to first date of study drug whether or not it was stopped before study drug administration.

[1] Medications were coded using WHO-DD (Enhanced version Sep. 2017), ATC Level 4

SOURCE: Listings xx.x.x, xx.x.x

Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311 Statistical Analysis Plan,



BlackThorn Therapeutics, Inc. Protocol NEP-PD-201 Table 14.2.1.1

FINAL 

Summary of UPDRS Part III Total Score pre-dose to post-dose on Day 1 Modified Intent-to-Treat Population

| Parameter | BTRX-246040 | BTRX-246040 | BTRX-246040 | Pooled | |
|---|---|---|---|---|---|
| Timepoint | 40 mg | 80 mg | 120 mg | BTRX-246040 | Placebo |
| Statistics | (N=XX) | (N=xx) | (N=xx) | (N=XX) | (N=xx) |
| LIPDRS Part III Total Score | | | | | |
| Pre-Dose Day 1 | | | | | |
| C | × | × | × | × | × |
| Mean (95% CI) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) |
| Standard Deviation | XX.XXX | XX.XX | XX.XXX | XX.XXX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum, Maximum | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xxx, xx.x | xx.x, xx.x |
| Post-Dose Day 1, <timepoint></timepoint> | | | | | |
| ٦ | × | ×× | XX | × | XX |
| Mean (95% CI) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) |
| Standard Deviation | XX.XXX | XX.XXX | XX.XXX | XX.XX | XX.XXX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum, Maximum | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

(Repeat for all post-dose timepoints, add descriptive summary for maximal change on Day 1 after all post dose day 1 timepoints summarized} Note: Treatment groups are based on treatment assigned.

SOURCE: Listings xx.x.x, xx.x.x

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY

Statistical Analysis Plan, Sponsor BlackThom Therapeutics Protocol Number NEP-PD-201 PCN Number 7311



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Table 14.2.1.2

Modified Intent-to-Treat Population AUC of UPDRS Part III Total Score

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | Pooled | |
|---|---|---|---|---|---|
| Parameter | 40 mg | 80 mg | 120 mg | BTRX-246040 | Placebo |
| Statistics | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| AUC | | | | | |
| u | × | X | × | XX | × |
| Mean (95% CI) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) |
| Standard Deviation | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum, Maximum | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X |

Note: Treatment groups are based on treatment assigned.

SOURCE: Listings xx.x.x, xx.x.x

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMIMMYYYY at HH:MM on data extracted on DDMIMMYYYY


 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Table 14.2.2

Summary of Dyskinesia Rating on Day 1 Modified Intent-to-Treat Population

| Parameter<br>Timepoint<br>Statistics | BTRX-246040<br>40 mg | BTRX-246040<br>80 mg | BTRX-246040<br>120 mg | Pooled<br>BTRX-246040 | Placebo |
|---|---|---|---|---|---|
| Dyskinesia Rating | (ox-a) | (SX-A) | (22-21) | (227-21) | (22-21) |
| Pre-Dose Day 1 | ; | ; | | ; | ; |
| 0 - No dyskinesia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx |
| 1 - Minimal or slight dyskinesia | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x:x%) xx |
| 2 - Mild dyskinesia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| 3 - Moderate dyskinesia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| 4 - Severe dyskinesia | (%x.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| Post-Dose Day 1, <timepoint></timepoint> | | | | | |
| 0 - No dyskinesia | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| 1 - Minimal or slight dyskinesia | xx (xx.x%) | (%x.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| 2 - Mild dyskinesia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| 3 - Moderate dyskinesia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| 4 - Severe dyskinesia | (%x.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| Post-Dose Day 1 Change, <timepoint></timepoint> | | | | | |
| u | XX | X | × | XX | × |
| Mean (95% CI) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) |
| Standard Deviation | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

## {Repeat for all post-dose timepoints}

Note: Percentages are 100\*n/N. Treatment groups are based on treatment assigned.

SOURCE: Listings xx.x.x, xx.x.x T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMIMMYYYY at HH:MM on data extracted on DDMIMMYYYY



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Table 14.2.3 Summary of Duration of ON and Time to ON on Day 1 Modified Intent-to-Treat Population

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | Pooled | |
|---|---|---|---|---|---|
| Parameter | 40 mg | 80 mg | 120 mg | BTRX-246040 | Placebo |
| Statistics | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Duration of ON, Day 1 (hours) | | | | | |
| L | × | × | × | XX | ×× |
| Mean (95% CI) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) |
| Standard Deviation | XX.XX | XX.XX | XX.XXX | XX.XX | XX.XXX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| Time to ON Part (house) | | | | | |
| IIIIIe to Oiv, Day I (IIOuis) | | | | | |
| u | × | × | × | × | ×× |
| Mean (95% CI) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) |
| Standard Deviation | XX.XX | XX.XX | XX.XXX | XX.XX | XX.XXX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Subjects that turn ON, Day 1 | (%x.xx) xx | (xx.x%) | (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Percentages are 100\*n/N. Treatment groups are based on treatment assigned. Duration of ON, Day 1 = First returned to OFF state datetime (UPDRS2 or DFUP CRF Page) - First reported ON state datetime (UPDRS2 CRF Page). Time to ON, Day 1 = First reported ON state datetime (UPDRS2 CRF Page) - Study drug administration datetime (EX1 CRF Page).

SOURCE: Listings xx.x.x, xx.x.x







Note: Treatment groups are based on treatment received.

SOURCE: Listings xx.x.x, xx.x.x T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY





 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Table 14.3.1.1
Summary of all AEs
Safety Population

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| | 40 mg | 80 mg | 120 mg | Placebo |
| Category | (N=xx) | (N=xx) | (N=XX) | (N=xx) |
| Subjects with at least one [1] | | | | |
| Treatment Emergent Adverse Event (TEAE) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | (%x.x%) | xx (xx.x%) | xx (xx.x%) |
| TEAE Potentially Related to Study Drug | (%x.x%) xx | xx (xx.x%) | (%x.xx) xx | (%x.x%) |
| Serious Adverse Event (SAE) | xx (xx.x%) | (%x.xx) xx | (%x.x%) | xx (xx.x%) |
| SAE Potentially Related to Study Drug | (%x.x%) xx | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) |
| Adverse Event Leading to Discontinuation | xx (xx.x%) | (%x.x%) | (%x.x%) | xx (xx.x%) |
| Adverse Event Leading to Death | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) |

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. Subjects were counted only once for each System Organ Class and Preferred Term. and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = related). TEAEs are defined as AEs Additionally, each subject is counted at the most once within the most severe event under the summary of severity TEAEs. If a particular event is missing the severity which start after the first dose of study medication.

[1] Adverse Events were coded using MedDRA version 20.1.

SOURCE: Listings xx.x.x, xx.x.x

Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311 Statistical Analysis Plan,



FINAL 

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

TEAEs by SOC, and Preferred Term Safety Population Table 14.3.1.2

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| System Organ Class [1] | 40 mg | 80 mg | 120 mg | Placebo |
| Preferred Term | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Number of subjects with at least one TEAE | (%* **) ** | (%^ ^x) *x | (%× ××) ×× | (%× ××) ×× |
| | (6/8:88) 88 | (6/2:22) 22 | (6/8:88) 88 | (6/2002) 22 |
| SOC 1 | xx (xx.x%) | xx (xx.x%) | (%x.x%) | (%x.x%) |
| PT 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| PT 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| PT3 | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx |
| SOC 2 | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| PT 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |

{Repeated for all applicable SOC/PT combinations}

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. Subjects were counted only once for each System Organ Class and Preferred Term. TEAEs are defined as AEs which start after the first dose of study medication.

[1] Adverse Events were coded using MedDRA version 20.1.

SOURCE: Listings xx.x.x, xx.x.x

Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311 Statistical Analysis Plan,



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201 Table 14.3.1.3

TEAEs by SOC, Preferred Term and Severity Safety Population

| System Organ Class [1] | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| Preferred Term | 40 mg | 80 mg | 120 mg | Placebo |
| Severity | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Number of subjects with at least one TEAE | xx (xx.x%) | xx (xx.x%) | (xx.x%) | (%x.xx) xx |
| | | Š | | |
| SOC 1 | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) |
| Mild | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| PT 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

# {Repeated for all applicable SOC/PT combinations}

under highest severity. If a particular event is missing the severity, then the strongest possible severity will be assumed for analysis (severity = severe). TEAEs are defined Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. Subjects were counted only once for each System Organ Class and Preferred Term as AEs which start after the first dose of study medication.

[1] Adverse Events were coded using MedDRA version 20.1.

SOURCE: Listings xx.x.x, xx.x.x



Table 14.3.1.4

TEAEs by SOC, Preferred Term and Relationship to Study Medication

Safety Population

{Programming Note: Repeat 14.3.1.3 with relationship to study medication levels and change Severity in the footnotes to Relationship. For the strongest possible relationship, put (relationship = related)}

Table 14.3.1.5

TEAEs leading to discontinuation by SOC and Preferred Term

Safety Population

{Programming Note: Repeat 14.3.1.2 subset to TEAEs leading to discontinuation}

Table 14.3.1.6

TESAEs other than deaths by SOC and Preferred Term

Safety Population

{Programming Note: Repeat 14.3.1.2 subset to TESAEs other than deaths}

Table 14.3.1.7

TEAEs leading to death by SOC and Preferred Term

Safety Population

{Programming Note: Repeat 14.3.1.2 subset to TEAEs leading to death}



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Table 14.3.2.1 Summary of Clinical Chemistry by Study Visit Safety Population

| Analyte | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| Visit | 40 mg | 80 mg | 120 mg | Placebo |
| Statistics | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Analyte (unit) | | | | |
| Baseline | | | | |
| u | ×× | × | ×× | ×× |
| Mean (95% CI) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) |
| Standard Deviation | XX.XX | XX.XXX | XX.XXX | xx.xx |
| Median | XX.XX | xx.xx | XX.XX | XX.XX |
| Minimum, Maximum | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Follow-up/ET | | | | |
| u | × | × | × | × |
| Mean (95% CI) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) | xx.xx (x.xx, x.xx) |
| Standard Deviation | XX.XX | XX.XXX | XX.XX | xx.xxx |
| Median | XX.XX | xx.xx | xx.xx | XX.XX |
| Minimum, Maximum | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |

{Programming Note: Continue for all applicable parameters, presenting change from baseline after the summary statistics for Follow-up/ET}

Note: Treatment groups are based on treatment received. The last non-missing observation recorded on or before the first dose of study drug will be used as the baseline observation.

SOURCE: Listings xx.x.x, xx.x.x



Table 14.3.2.2 Summary of Hematology by Study Visit Safety Population

{Programming Note: Repeat 14.3.2.1 with hematology analytes}

Table 14.3.2.3 Summary of Urinalysis by Study Visit Safety Population

{Programming Note: Repeat 14.3.2.1 with urinalysis analytes}

Table 14.3.2.4
Summary of Coagulation by Study Visit
Safety Population
{Programming Note: Repeat 14.3.2.1 with coagulation analytes}



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Table 14.3.2.5 Shifts from Baseline of Clinical Chemistry by Study Visit Safety Population

| | | | | | | Base | Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | - | BTRX-246040 | 0 | Ш | BTRX-246040 | | - | BTRX-246040 | | | | |
| Analyte | | 40 mg | | | 80 mg | | | 120 mg | | | Placebo | |
| Follow-up/ET Results | | (N=xx) | | | (N=xx) | | | (N=xx) | | | (N=xx) | |
| | Low | Normal | High | Low | Normal | High | Low | Normal | High | Low | Normal | High |
| Analyte (unit) | | | | | | | | | | | | |
| Low | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx (%x.x%) xx (xx.x%) xx (%x.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) |
| Normal | (%x.x%) | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx |
| High | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.x%) xx (%x.x%) xx (%x.x%) xx | xx (xx.x%) | xx (xx.x%) | (%x.x%) xx | xx (xx.x%) | xx (xx.x%) |
| Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) xx (xx.x%) | xx (xx.x%) | (%x.x%) xx (%x.x%) xx (%x.x%) xx (%x.x%) xx | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) xx (xx.x%) | xx (xx.x%) |
| Analyte (unit) | | | | | | | | | | | | |
| Low | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | (2,000) XX (3,000) XX | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) |
| Normal | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx (%x.x%) xx (%x.x%) xx (%x.x%) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx (%x.xx) xx | (%x.xx) xx |
| High | (%x.x%) xx | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | (%x.x%) xx | xx (xx.x%) | xx (xx.x%) xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) |
| Missing | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | (%x.x%) xx (%x.x%) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) xx (xx.x%) xx (xx.x%) xx | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx (%x.xx) xx (%x.xx) xx | (%x.xx) xx | (%x.xx) xx |

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. Baseline result is presented horizontally across the top, and Follow-up/ET result is presented vertically in the first column. The last non-missing observation recorded on or before the first dose of study drug will be used as the baseline observation. SOURCE: Listings xx.x.x, xx.x.x



Table 14.3.2.6

Shifts from Baseline of Hematology by Study Visit

Safety Population

{Programming Note: Repeat 14.3.2.4 with hematology analytes}

Table 14.3.2.7

Shifts from Baseline of Urinalysis by Study Visit Safety Population

{Programming Note: Repeat 14.3.2.4 with urinalysis analytes}

Table 14.3.2.8

Shifts from Baseline of Coagulation by Study Visit

Safety Population

{Programming Note: Repeat 14.3.2.4 with coagulation analytes}

Table 14.3.3.1

Summary of Vital Signs by Study Visit

Safety Population

{Programming Note: Repeat 14.3.2.1 with vital signs parameters and all applicable study visits/change from baselines}

Table 14.3.3.2

Summary of Orthostatic Blood Pressure and Pulse by Study Visit

Safety Population

{Programming Note: Repeat 14.3.2.1 with orthostatic blood pressure and pulse for all applicable study visits/change from baselines. The Average of the three BP and Pulse measurements will be used for baseline, update footnote as applicable (as in 14.3.3.3) to reflect this}

Version 1.1 | Date 23-Sep-2019 | AD-PR-109.01 Effective date: 26-Jun-2017

Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311 Statistical Analysis Plan,



FINAL 

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Incidence of Abnormal Orthostatic Blood Pressure by Study Visit Safety Population Table 14.3.3.3

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| Visit | 40 mg | 80 mg | 120 mg | Placebo |
| Change from Baseline | (N=XX) | (N=xx) | (N=XX) | (N=xx) |
| Day 1 2 hours nost-dosa | > | } | > | > |
| שלא אלי ביוסמים שליים שלים של | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | XX | XX XX |
| >= 20 mmHg systolic blood pressure drop | (%x.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| >= 10 mmHg diastolic blood pressure drop | (%x.x%) xx | xx (xx.x%) | (%x.x%) | (%x.x%) |
| Day 1, 4 hours post-dose | × | × | × | × |
| >= 20 mmHg systolic blood pressure drop | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| >= 10 mmHg diastolic blood pressure drop | (%x.x%) | (%x.x%) xx | xx (xx.x%) | xx (xx.x%) |
| Day 1, 6 hours post-dose | ×× | × | × | × |
| >= 20 mmHg systolic blood pressure drop | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| >= 10 mmHg diastolic blood pressure drop | (%x.x%) xx | (%x.x%) | xx (xx.x%) | (%x.xx) xx |
| Day 1, 8 hours post-dose | X | × | × | × |
| >= 20 mmHg systolic blood pressure drop | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| >= 10 mmHg diastolic blood pressure drop | (%x.x%) xx | (%x.x%) | xx (xx.x%) | xx (xx.x%) |
| Follow-up/ET | X | × | × | × |
| >= 20 mmHg systolic blood pressure drop | xx (xx.x%) | xx (xx.x%) | (%x.x%) | xx (xx.x%) |
| >= 10 mmHg diastolic blood pressure drop | x (xx.x%) | (%x.x%) | xx (xx.x%) | xx (xx.x%) |

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. The average of the three BP and pulse measurements will be used for comparison to all post-treatment measurements to minimize the impact of biological variability and to serve as a more reliable baseline orthostatic vital sign measurement..

SOURCE: Listings xx.x.x, xx.x.x TS\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY



Summary of ECG Parameters by Study Visit Safety Population Table 14.3.3.4

{Programming Note: Repeat 14.3.2.1 with ECG parameters and all applicable study visits/change from baselines}



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Incidence of Abnormal ECG by Study Visit Safety Population Table 14.3.3.5

| | BTRX-246040 | BTRX-246040 | BTRX-246040 | |
|---|---|---|---|---|
| Visit | 40 mg | 80 mg | 120 mg | Placebo |
| Category | (N=XX) | (N=xx) | (N=XX) | (N=xx) |
| Baseline | × | XX | × | × |
| Normal | (%x.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal, not clinically significant | xx (xx.x%) | (%x:x%) | xx (xx.x%) | (%x.xx) xx |
| Abnormal, clinically significant | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| Day 1, 1 hour post-dose | × | XX | × | × |
| Normal | xx (xx.x%) | xx (xx.x%) | (%x.x%) | (%x.x%) |
| Abnormal, not clinically significant | xx (xx.x%) | (%x:x%) | xx (xx.x%) | (%x.x%) |
| Abnormal, clinically significant | xx (xx.x%) | (%x.x%) | xx (xx.x%) | (%x.x%) xx |
| Follow-up/ET | × | XX | × | × |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal, not clinically significant | (%x.x%) | xx (xx.x%) | xx (xx.x%) | (%x.x%) |
| Abnormal, clinically significant | (%x.x%) | xx (xx.x%) | xx (xx.x%) | (%x.x%) |

Note: Percentages are 100\*n/N. Treatment groups are based on treatment received. The last non-missing observation recorded on or before the first dose of study drug will be used as the baseline observation.

SOURCE: Listings xx.x.x, xx.x.x T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY



Table 14.3.4.1 Summary of Impulsive Control Disorder and QUIP-RS by Study Visit

{Programming Note: Repeat 14.3.2.1 with QUIP-RS and Impulsive Control Disorder parameters (including Total ICD, Total QUIP-RS) and all applicable study visits/change from baselines} Safety Population



#### 12.3. Planned Figure Shells

Figure 14.2.1 AUC of UPDRS Part III Total Score

Modified Intent-to-Treat Population

(Programming Note: Line plot by cohort for 8 hours of collected UPDRS Part III Total Scores. Y = UPDRS Part III Score, X = Time

Figure 14.2.2

Scatter Plot of maximal change in UPDRS Part III Total Score

Modified Intent-to-Treat Population

{Programming Note: Scatter plot by cohort of maximum change for UPDRS Part III Total Scores. Y = Change in UPDRS Part III Score, X = Time}

Figure 14.2.3

Scatter Plot of UPDRS Part III Total Score by timepoint

Modified Intent-to-Treat Population

{Programming Note: Scatter plot by cohort of UPDRS Part III Total Scores. Y = UPDRS Part III Score, X = Individual Timepoints}

Figure 14.3.1

Scatter Plot of serum concentration (linear)

Safety Population

{Programming Note: Scatter plot by cohort of serum concentration (active treatment only). Y = serum concentration (linear scale), X = Time}

Figure 14.3.2

Scatter Plot of serum concentration (logarithmic)

Safety Population

{Programming Note: Scatter plot by cohort of serum concentration (active treatment only). Y = serum concentration (log scale), X = Time}



### 12.4. Planned Listing Shells

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Listing 16.2.1.1
Assignment to Analysis Populations and Treatment Arm All Subjects Screened

 FINAL

| SAF | Yes | Yes | Yes | N<br>O |
|---|---|---|---|---|
| тIш | Yes | Yes | Yes | No |
| Treatment | XXXXXX | XXXXXXXXX | XXXXXX | |
| Treatment | XXXXXX | XXXXXXXXX | XXXXXX | |
| Cohort | Cohort 1 | Cohort 2 | Cohort 3 | |
| Number | XXX | XXX | XXXX | |
| Date | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | |
| Randomized? | Yes | Yes | Yes | ON. |
| Subject ID | XXXX | XXXXX | XXXX | XXXXX |
| | Randomized? Date Number Cohort Treatment Treatment mITT | Randomized? Date Number Cohort Treatment mITT Yes DDMIMMYYYY XXXX Cohort 1 xxxxxxx xxxxxx Yes | Randomized? Date Number Cohort Treatment mITT Yes DDMIMMYYYY XXXX Cohort 1 xxxxxxxx Yes Yes DDMIMMYYYY XXXX Cohort 2 xxxxxxxxx Xxxxxxxx Yes | Randomized? Date Number Cohort Treatment Treatment mITT Yes DDMIMMYYYY XXXX Cohort 1 xxxxxxxxx Yes Yes DDMIMMYYYY XXXX Cohort 2 xxxxxxxxx Yes |

Note: mITT = Modified Intent-to-Treat Population, SAF = Safety Population. T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMIMMYYYY at HH:MM on data extracted on DDMIMMYYYY



BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Listing 16.2.1.2

 FINAL

> Study Completion Status and Reasons for Discontinuation All Subjects Screened

> > Planned Treatment: XXXXXXX

| Subject ID | Subject ID Screen Date | Completed<br>Study? | Date<br>Completed | Date of<br>Discontinuation | Reason for<br>Discontinuation | Date of Last<br>Contact if Lost to<br>Follow-Up/<br>Reason | Date of Death/<br>Reason | Was the Blind Broken for this<br>Subject?/<br>Date Broken/<br>Reason |
|---|---|---|---|---|---|---|---|---|
| XXXXX | DDMMMYYYY | Yes | DDMMMYYYY | | | DDMMMYYYY | | |
| XXXXX | DDMMMYYYY | Yes | DDMMMYYYY | DDMMMYYYY | XXXXXXXXXX | DDMIMIMYYYY/<br>xxxxxx xxxx | DDMMMYYYY/<br>xxxxxxxxx | Yes/ DDMIMMYYYY/<br>xxxxxxxx xxxx x xxxxxx xxxx |
| XXXX | DDMMMYYYY | ON. | | DDMMMYYYY | XXXXXXXXXX | DDMMMYYYY | | |
| XXXXX | DDMMMYYYY | Yes | DDMMMYYYY | | | DDMMMYYYY | | |

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMIMMYYYY at HH:MM on data extracted on DDMIMMYYYY

randomization discontinuations, put NCOMPLT. In addition, for AE, PHYSICIAN DECISION, or OTHER, add a colon, a space, and the associated WITHDRAWAL OF CONSENT, ADVERSE EVENT, or OTHER: ). In the case of Other, also concatenate the Other specify reason. For post-{Programming Note: In the case of screen failure, put "SCREEN FAILURE," concatenated SCR\_FAIL.DSREAS (either ELIGIBILITY, specify reason.}



FINAL 

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Listing 16.2.1.3

Inclusion and Exclusion Criteria All Subjects Screened

| Description of Criteria Not Met | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | XXXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|---|
| Criteria Not Met | Inclusion #1, Exclusion #2 | | | Inclusion #9 |
| Did subject meet all eligibility<br>criteria? | ON | Yes | Yes | No |
| Subject ID | XXXXX | XXXXX | XXXXX | XXXXX |




BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Protocol Deviations Modified Intent-to-Treat Population Listing 16.2.2.1

| | | Event Category Description | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ************************************** | | | Αλλάλλλάλλλάλλ | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Major | Minor | 2 | NA: | _ | 20.00 |
| | Event | Subject ID Event Date Report Date Event Type | | DDMMMYYYY | NAMWAYYY | | | | |
| Planned Treatment: XXXXXXX | | <b>Event Date</b> | | DDMMMYYYY DDMMMYYYY | VVVVWWMMUU VVVVWMMMUU | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | NAME OF THE OWNER OF THE OWNER OF THE OWNER OF THE OWNER OWN |
| Planned Treat | | Subject ID | : | XXXXX | XXXX | XXXXXX | **** | <b>/////</b> | **** |



FINAL 

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Listing 16.2.4.1

Demographics Safety Population

| Actual Treatr | Actual Treatment: XXXXXXX | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Baseline | Baseline | Baseline |
| | Informed | | | | | | Years of | Weight | Height | BMI |
| Subject ID | Consent Date | Subject ID Consent Date Date of Birth Age (yrs) | Age (yrs) | Gender | Ethnicity | Race | Education | (kg) | (cm) | (kg/m2) |
| XXXXX | WWWW | XXXXMMMQQ XXXXMMMQQ | \$ | Female | ****** | ****** | \$ | > | \$ | ** |
| YYYYYY | | | ¥ | 5 | *************************************** | VVVVVVVVVV | ŧ. | V:VV | ¥ | VV:VV |
| XXXXX | DDMMMYYYY | ррмммүүүү ррмммүүү | × | Male | XXXXXXX | XXXXX | × | XX.X | × | XX.XX |
| XXXX | DDMMMYYYY | ррмимуүүү ррмммүүүү | × | Male | XXXXX | XXXX | × | XX.X | × | XX.XX |
| XXXXX | DDMMMYYYY | ррмимуүүү ррмммүүү | × | Female | XXXXXXXXX | xxxxxxxx | × | XX.X | × | XX.XX |



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Listing 16.2.4.2 Medical and PD History Safety Population

| Actual Treatment: XXXXXXX | System Organ Class [1]/ Preferred Term/ Start Date/ Medication given?/ Parkinson's Disease History Any History? Ongoing? Verbatim Term End Date Intensity Date of Diagnosis | Yes No XXXXXXXXXXXXXXXXX DDMMMYYYY No/xxxxX XXXXXXXX DDMMMYYYY DDMMMYYYY XXXXXXXXXX | Yes XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | No | Yes No XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|---|---|
| nent: XXXXXXX | | Yes | | NO | Yes |
| Actual Treatn | Subject ID | XXXX | XXXX | XXXXX | XXXXX |

<sup>[1]</sup> Medical history was coded using MedDRA version 20.1. T:\BlackThorn\ NEP-PD-201\..\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Listing 16.2.4.3
Concomitant and Prior Medications
Safety Population

Actual Treatment: XXXXXXX

| ערנממו וורמנוו | Actual II carillelle, MMMMM | | | | | |
|---|---|---|---|---|---|---|
| | | | Anatomic Therapeutic Class (level 4) [2]/ | | | Dose (unit)/ |
| | | | Preferred Term/ | Start Date (Study Day)/ | | Route/ |
| Subject ID | Any Meds? | Type [1] | Verbatim Term | End Date (Study Day) [3] | Indication | Frequency |
| XXXXX | Yes | O | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx) | XXXXXXXXX | XXXXXXXXXXXXXXXX <units> / XXXXXXX/ XXXXXXXXXXXXXXXXXXXXXXXXXXX</units> |
| | | U | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (xx)/<br>ONGOING | ×××××× | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXX | N<br>O | | | | | |
| XXXXX | Yes | ۵ | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY (xx)/<br>ONGOING | ×××××× | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

<sup>[1]</sup> C = Concomitant medication, administered during participation in the study, on or after first date of study drug; P = Prior Medication, administered prior to first date of study drug whether or not stopped prior to study drug administration.

<sup>[2]</sup> Medications were coded using WHO-DD Enhanced Version Sep. 2017, ATC level 4.

<sup>[3]</sup> Study Day = Assessment Date – Date of First Dose + 1

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY





FINAL 

BlackThorn Therapeutics, Inc.

Protocol NEP-PD-201

Listing 16.2.5.1.1

Drug Accountability Safety Population

| Planned Trea | Planned Treatment: XXXXXXX | | | | | | |
|---|---|---|---|---|---|---|---|
| | Drug | | | Bottle 1 dispensed/ | Bottle 2 dispensed/ | Bottle 1 dispensed/ Bottle 2 dispensed/ Bottle 3 dispensed/ Bottle 4 dispensed/ | Bottle 4 dispensed/ |
| Subject ID | Subject ID dispensed? | Reason not dispensed | Date dispensed | Bottle number | Bottle number | Bottle number | Bottle number |
| XXXXX | Yes | | DDMMMYYYY | Yes/xxxx | Yes/xxxx* | Yes/xxxx | Yes/xxxx |
| XXXXX | No | XXXXXXXXX XXXX | | | | | |
| XXXXX | Yes | | DDMMMYYYY | Yes/xxxx | Yes/xxxx | No | No |
| XXXXX | Yes | | DDMMMYYYY | Yes/xxx | Yes/xxxx | No | No |

{Programming Note: Bottle 4 dispensed date may not be necessary, please check data prior to including this column.}

<sup>\*</sup> Actual Treatment does not match Planned Treatment.

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY



 FINAL

BlackThorn Therapeutics, Inc.

Protocol NEP-PD-201

Listing 16.2.5.1.2 Study Drug Administration Safety Population

Stu

| | ules taken | | | | |
|---|---|---|---|---|---|
| | Number of capsules taken | XX | | × | × |
| | Time of administration | MH:MM | | HH:MM | HH:MM |
| | Date of administration | DDMMMYYYY | | DDMMMYYYY | DDMMMYYYY |
| | Reason not administered | | xxxxxxxxxx | | |
| Actual Treatment: XXXXXXX | Drug<br>Subject ID Administered? | Yes | No | Yes | Yes |
| Actual Treatr | Subject ID | XXXXX | XXXXX | XXXXX | XXXXX |





| <br>FINAL | Serum concentration (unit) | XX.XX<br>XX.XX<br>XX.XX<br>XX.XX |
|---|---|---|
| | Time collected | HH:MM<br>HH:MM<br>HH:MM<br>HH:MM |
| 040 | Date collected | DDMIMMYYYY<br>DDMIMMYYYY<br>DDMIMMYYYY<br>DDMIMMYYYY |
| Listing 16.2.5.2<br>Serum Concentration of BTRX-246040<br>Safety Population | Timepoint | Pre-dose 30 minutes post-dose 60 minutes post-dose 120 minutes post-dose 240 minutes post-dose 480 minutes post-dose |
| | Reason not collected | XXXXXXXXXXXX |
| b-201 D-xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Sample collected? | Ves<br>No<br>No<br>Res<br>No |
| BlackThorn Therapeutics, Inc. Protocol NEP-PD-201 Actual Treatment: XXXXXXX | Subject ID | XXXXX |

Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311 Statistical Analysis Plan,




BlackThorn Therapeutics, Inc. Protocol NEP-PD-201 Listing 16.2.6.1

Unified Parkinson's Disease Rating Scale (Part III) Modified Intent-to-Treat Population

| | | | Result | XXX | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | | XXX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Question Text | XXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | XXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX XXXXXXXXXX XXXXXXXX | <br>XXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | XXXXXXXXX XXXXXXXXXX XXXXXXXX |
| | | | Status | NO | | | | | | | | OFF | | |
| | | | Timepoint | 30 minutes | post-dose | | | | | | | 60 minutes | post-dose | |
| | | | Start time | HH:MM | | | | | | | | | | |
| | | Date of | Assessment | DDMMMYYYY | | | | | | | | | | |
| | | Reason not | completed | | | | | | | | | | | |
| Planned Treatment: XXXXXXX | Was | assessment | completed? | Yes | | | | | | | | | | |
| Planned Trea | | | Subject ID | XXXXX | | | | | | | | | | |

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY

{Programming Note: Dyskinesia rating and Total Score for UPDRS appears in 16.2.6.2, include screening UPDRS results, if more space is required combine time and date columns}



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Total UPDRS Score (Part III) and Dyskinesia Rating Modified Intent-to-Treat Population Listing 16.2.6.2

| | | Total UPDRS Score | nepoint Status (Part III) Dyskinesia Rating | į | 30 minutes ON xxx | post-dose | 60 minutes ON xxx xxxxxxxxxx | post-dose | 90 minutes ON xxx xxxxxxxxx | post-dose | .20 minutes ON xxx xxxxxxxxxx | post-dose |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Reason not Date of | completed Assessment Start time Timepoint Status | | DDMMMYYYY HH:MM | | | | | | | |
| Planned Treatment: XXXXXXX | Was | assessment R | Subject ID completed? c | | XXXXX Yes | | | | | | | |

T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY

{Programming Note: Include screening UPDRS results}



 FINAL

BlackThorn Therapeutics, Inc.

Protocol NEP-PD-201

Listing 16.2.6.3
Time to and Duration of ON state
Modified Intent-to-Treat Population

Planned Treatment: XXXXXXX

| | Duration of ON State (hrs) [2] | XXX.X | XXXXX | xxxx.x | xxxx.x |
|---|---|---|---|---|---|
| | Time to On State (hrs) [1] Dura | XXX.X | XXXX.X | XXX.X | XXX.X |
| | Study administration<br>Datetime | DDMMMYYYY: | DDMMMYYY:<br>HH:MM | ррмммүүүү:<br>НН:ММ | ррмммүүү:<br>нн:мм |
| | Off State<br>Datetime | DDMMMYYYY: | DDMMIMYYYY:<br>HH:MM | DDMMMYYYY:<br>HH:MM | БРМММҮҮҮҮ:<br>НН:ММ |
| Planned Treatment: XXXXXXX | On State<br>Datetime | DDIMMIMYYYY: | DDMMMYYYY:<br>HH:MM | ррмммүүүү:<br>нн:мм | ррмммүүүү:<br>нн:мм |
| Planned I reatm | Subject ID | XXXXX | ×××× | XXXXX | XXXXX |

<sup>[1]</sup> Duration of ON time on Day 1 = First returned to OFF state Datetime (UPDRS2 or DFUP CRF Page) - First reported ON state Datetime (UPDRS2 CRF Page). [2] Time to ON on Day 1 = First reported ON state Datetime (UPDRS2 CRF Page) - Study drug administration Datetime (EX1 CRF Page) T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMIMMYYYY at HH:MM on data extracted on DDMMIMYYYY



FINAL


BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Listing 16.2.7.1
Treatment-emergent adverse events
Safety Population

Actual Treatment: XXXXXXX

| CA/DIS/HO/<br>DE/LT/OTH [4] | /oN/oN/oN<br>No/No/No | No/No/Yes/<br>No/No/Yes | No/No/No/<br>No/No/No |
|---|---|---|---|
| Serious | o<br>Z | Yes | <u>8</u> |
| Outcome/<br>Study Med<br>Action<br>Taken/Other<br>Action Taken | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | /xxxxxxxxxxx/<br>/xxxxxxxxxxxxxxxxxxxxxxx | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| Severity/<br>Relationship to<br>Study Drug | xxxxxxx/<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| Event Duration<br>(days:hrs:min) [3] | DD:HH:MM | рр:нн:мм | DD:HH:MM |
| Start Datetime (Study Day) [2]/<br>End Datetime (Study Day) | БРМММҮҮҮҮ:НН:ММ (xx)/<br>БРМММҮҮҮҮ:НН:ММ (xx) | DDMMMYYYY:HH:MM (xx)/<br>DDMMMYYYY:HH:MM (xx) | DDMIMMYYYY:HH:MM (xx)/<br>ONGOING |
| System Organ Class [1]/<br>Preferred Term/<br>Verbatim Term | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXX |
| Subject ID | XXXX | XXXX | XXXX |

<sup>[1]</sup> Adverse Events were coded using MedDRA version 20.1.

{Programming Note: Event duration will be displayed as DD:HH:MM, and is the difference of end datetime – start datetime + 1. if other action is populated, concatenate with action taken with study medication separated by semi-colon. If there is "Procedure, specify" or "Other, specify" details, they would also need to be presented here. If Death is marked as Yes, add date in column for death date pulled from disposition data separated by semi-colon. }

<sup>[2]</sup> Study Day = Assessment Date – Date of First Dose + 1.

<sup>[3]</sup> Days:Hours:Minutes is based on End Date & Time – Start Date & Time + 1

<sup>[4]</sup> CA = Congenital abnormality or birth defect, DE = Death (fatal), DIS = Persistent or significant disability/incapacity, HO = Hospitalization or prolongation of hospitalization, LT = Life-threatening event, OTH = Other important medical event.

T.\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY



Listing 16.2.7.2
Serious adverse events
Safety Population

Safety Population {Programming Note: Repeat 16.2.7.1 with only SAEs}

Listing 16.2.7.3 Adverse Events leading to discontinuation

Safety Population {Programming Note: Repeat 16.2.7.1 with only AEs leading to discontinuation}

Listing 16.2.7.4 Listing of deaths Safety Population

Safety Population {Programming Note: Repeat 16.2.7.1 with only fatal AEs}

Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311 Statistical Analysis Plan,



FINAL 

BlackThorn Therapeutics, Inc.

Protocol NEP-PD-201

Clinical Chemistry Safety Population Listing 16.2.8.1

| | | | | | Accession Number | XXXXXXX | | | XXXXXXXXX | | XXXXXXX | | XXXXXXXX | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Change from Baseline | | | | XXX | | | | XXX | |
| | Standard | Reference | Range | | High | × | | | × | | × | | × | |
| | Stan | Refer | Rar | | Low | × | | | × | | × | | × | |
| | | | | | Units | XXXX | | | XXXXX | | XXXXX | | XXXXX | |
| | | | Test | Result | [2] | XXXX | | | ×xxxxx | | XXXXX | | XXXXX | |
| | | | | Sample | collected? | Yes | No | | Yes | | Yes | | Yes | |
| | | | | Collection Date/ | Collection Time | DDMMMYYYY/ | DDMMMYYYY/ | HH:MM | DDMMMYYYY/ | HH:MM | DDMMMYYYY/ | HH:MM | DDMMMYYYY/ | HH:MM |
| | | | Visit | (Study | Day[1]) | (xx) xxx | (xx) xxx | | (xx) xxx | | (xx) xxx | | (xx) xxx | |
| ent: XXXXXXX | | | | Analyte | (units) | XXXXXXXX | | | | | XXXXXXXXX | | | |
| Actual Treatment: XXXXXXX | | | | Subject ID | /Age/Sex | XXXXXXXX M/XX/XXXXX | | | | | XXXXX/XX/F | | | |

<sup>[1]</sup> Study Day = Assessment Date - Date of First Dose + 1

<sup>[2]</sup> L = low result, H = high result, ^ = abnormal result. T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMIMMYYYY

<sup>(</sup>Programming note, if abnormal, add clinical significance if collected to test result column)



Listing 16.2.8.2 Hematology

Safety Population

{Programming Note: Repeat 16.2.8.1 with hematology analytes}

Safety Population Listing 16.2.8.3 Urinalysis

{Programming Note: Repeat 16.2.8.1 with urinalysis analytes}

Listing 16.2.8.4

Coagulation
Safety Population
{Programming Note: Repeat 16.2.8.1 with coagulation analytes}



 FINAL

BlackThorn Therapeutics, Inc.

Protocol NEP-PD-201

Urine Drug Screen Safety Population Listing 16.2.8.5

Actual Treatment: XXXXXX

| Comments | | XXXXXX | | | XXXXXXX | XXXXXX | XXXXXXX | | |
|---|---|---|---|---|---|---|---|---|---|
| Test Result<br>[2] | XXXXX | | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| Reason not<br>Performed | | XXXXXXXXX | | | | | | | |
| Drug Screen Performed? | Yes | No | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| Date and Time Performed | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM |
| Visit<br>(Study Day[1]) | (xx) xxx | (xx) xxx | (xx) xxx | (xx) xxx | (xx) xxx | (xx) xxx | (xx) xxx | (xx) xxx | (xx) xxx |
| Analyte | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX |
| Subject ID | XXXXX | | | | | | | | |

[1] Study Day = Assessment Date — Date of First Dose + 1 T:\BlackThorn\\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY



 FINAL

BlackThorn Therapeutics, Inc.

Protocol NEP-PD-201

Actual Treatment: XXXXXXX

Safety Population Listing 16.2.9.1 Vital Signs

| Diastolic | BIOOG | Pressure | (mmHg) | | | | ××× | | ××× | | | ××× | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Systolic | B1000 | Pressure | (mmHg) | | | | ××× | | ××× | | | XXX | | | |
| | | Pulse | (beats/min) | | | | XXX | | XXX | | | XXX | | | |
| | Kespir- | ation Rate | (pbm) | | | | XXX | | XXX | | | XXX | | | |
| | | Temp | (C) | | XXX.X | | | | | | XXX.X | | | | |
| 2 | 2 | (kg/ | m2) | | XX.X | | | | | | XX.X | | | | |
| | | Weight | | | XXX.X | | | | | | XXX.X | | | | |
| | | Height | (cm) | | XXX.X | | | | | | x.xx.x | | | | |
| 9 | Keason | not | collected | | | | | | | | | | | XXXXXX | |
| | | Vital Signs | Collected? | 7 | Yes | | Yes | | Yes | | Yes | Yes | | N <sub>o</sub> | |
| | | Datetime of | Measurement | | DDIMIMINAYYY: | HH:MM | DDMMMYYYY: | HH:MM | DDMMMYYYY: | HH:MM | DDMMMYYYY | DDMMMYYYY: | HH:MM | DDMMMYYYY: | HH:MM |
| | | | Position | ×, | N/A | | Supine | | Standing | | N/A | Supine | | Standing | |
| #:0:// | VISIT | (Study | Day[1]) | | (xx) xxx | | (xx) xxx | | (xx) xxx | | (xx) xxx | (xx) xxx | | (xx) xxx | |
| | | | Subject ID Day[1]) | 20000 | XXXXX | | | | | | | | | | |

<sup>[1]</sup> Study Day = Assessment Date – Date of First Dose + 1 T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY



 FINAL

BlackThorn Therapeutics, Inc.

Protocol NEP-PD-201

Electrocardiogram Safety Population Listing 16.2.9.2

Actual Treatment: XXXXXXX

| Investigator<br>Interpretation<br>[2] | Normal<br>Normal | Normal<br>Abnormal, NCS | Abnormal, NCS |
|---|---|---|---|
| RR<br>(msec) | × ×<br>× × | × ×<br>× × | ×× |
| QTcF<br>(msec) | XX XX | XX XX | XXX |
| QTcB<br>(msec) | × × × | × × × | × |
| QT<br>(msec) | ××× | ××× | ××× |
| QRS<br>(msec) | ××× | ××× | ××× |
| PR<br>(msec) | ××× | × ×<br>× × | ×× |
| Reason<br>not<br>collected | | | ××××× |
| ECG<br>Collected? | Yes<br>Yes | Yes<br>Yes | No<br>Yes |
| Time | ∑ | Σ Σ<br>Σ Σ<br>Ε Η Η<br>Η Η | ∑ |
| Date of<br>Measurement | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY |
| Visit<br>(Study<br>Day[1]) | (xx) xxx | (xx) xxx | (xx) xxx |
| Visit (Study Subject ID Day[1]) | XXXX | XXXX | XXXX |

<sup>[1]</sup> Study Day = Assessment Date - Date of First Dose + 1

<sup>[2]</sup> CS = clinically significant, NCS = not clinically significant. T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMIMMYYYY

Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311 Statistical Analysis Plan,



FINAL 

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Physical Examination Safety Population Listing 16.2.9.3

Actual Treatment: XXXXXXX

| Clinically<br>Significant [2] | NCS | S |
|---|---|---|
| Abnormal<br>Findings | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXXX |
| Result | XXXXXXXXXX XXXX XXXXXXXXX XXXXXXXXX | XXXXXXXXX |
| Body System | XXXXXXX<br>XXXXXXX<br>XXXXXXX<br>XXXXXXX<br>XXXXXXX | XXXXXX |
| Performed? | Yes | |
| Exam | Ж.<br>Ж. | |
| Exam Date | ррмммүүү | |
| Visit<br>(Study<br>Day[1]) | (xx) xxx | |
| Visit<br>(Study<br>Subject ID Day[1]) | XXXXX | |

<sup>[1]</sup> Study Day = Assessment Date - Date of First Dose + 1

Neurological Examination Listing 16.2.9.4

Safety Population [Programming Note: Repeat 16.2.9.3, use applicable Neurological Examination question text/results. In the header, replace "Body System" with "Neurological System" [Programming Note: Repeat 16.2.9.3, use applicable Neurological Examination question text/results.]

<sup>[2]</sup> CS = clinically significant, NCS = not clinically significant. T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMIMMYYYY



Listing 16.2.9.5

Columbia-Suicide Severity Rating Scale (C-SSRS)

Safety Population

{Programming Note: Repeat 16.2.6.1, drop timepoint, status and use applicable C-SSRS question text/results}

Listing 16.2.9.6

Questionnaire for Impulsive-Compulsive Disorders in Parkinson's disease Rating Scale (QUIP-RS)

Safety Population

{Programming Note: Repeat 16.2.6.1, drop timepoint, status and use applicable QUIP-RS question text/results, including ICD, QUIP-RS}

Version 1.1 | Date 23-Sep-2019 | AD-PR-109.01 Effective date: 26-Jun-2017

Sponsor BlackThorn Therapeutics Protocol Number NEP-PD-201 PCN Number 7311 Statistical Analysis Plan,



BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Montreal Cognitive Assessment (MoCA) Safety Population Listing 16.2.9.7

FINAL 

Actual Treatment: XXXXXXX

| Total | ××× | × ×<br>× × | ×× |
|---|---|---|---|
| 08 | ×× | ž ž | × |
| Ω7 | ×× | ×× | × |
| 96 | ×× | ×× | × |
| | ×× | ×× | × |
| Q4 Q5 | ×× | ×× | × |
| 03 | ×× | ×× | × |
| 02 | ×× | ×× | × |
| 0,1 | ×× | ×× | × |
| Reason<br>not<br>collected | | | ××××× |
| Assessment<br>Collected? | Yes | Yes | No<br>Yes |
| Time<br>Collected | M M M M M M M M M M M M M M M M M M M | ΣΣ | ΣΣ |
| Time<br>Collecte | ΗΉ | HH:MM:HH:MM | M:HH<br>H:MM |
| Date of Tir<br>Assessment Colle | DDMMMYYYY HH: | DDMMMYYYY HH:M<br>DDMMMYYYY HH:M | DDMMMYYYY HH:M<br>DDMMMYYYY HH:M |

Note: Q1 = Visuospatial/Executive, Q2 = Naming, Q3 = Memory, Q4 = Attention, Q5 = Language, Q6 = Abstraction, Q7 = Delayed Recall, Q8 = Orientation [1] \* = Subject has less than or equal to 12 years of education. For these subjects, 1 point is added to the total score.

<sup>[2]</sup> Study Day = Assessment Date – Date of First Dose + 1 T:\BlackThorn\ NEP-PD-201\...\xxxxxx.sas run on DDMMMYYYY at HH:MM on data extracted on DDMMMYYYY



Listing 16.2.9.8
Beck Depression Inventory-II

Safety Population (Programming Note: Repeat 16.2.9.7, update footnote and stack columns as necessary to fit additional questions)



 FINAL

BlackThorn Therapeutics, Inc. Protocol NEP-PD-201

Listing 16.2.9.9 Modified Hoehn and Yahr scale Safety Population

Actual Treatment: XXXXXXX

| Hoehn and Yahr Staging Score | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX |
|---|---|---|---|
| Time<br>Collected | HH:MM<br>HH:MM | HH:MM<br>HH:MM | HH:MM |
| Date of Assessment | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY |
| Visit<br>(Study<br>Day[1]) | (xx) xxx | (xx) xxx | (xx) xxx |
| Visit (Study Subject ID Day[1]) | XXXX | XXXX | XXXX |

[1] Study Day = Assessment Date – Date of First Dose + 1





#### **Appendix 1: Library of Abbreviations**

| Abbreviation | Definition |
|--------------|----------------------------------------|
| ATC | anatomical therapeutic chemical |
| AUC | area under the curve |
| BLQ | beneath limit of quantification |
| BMI | body mass index |
| CI | confidence interval |
| CRF | case report form |
| CRO | contract research organization |
| CS | clinically significant |
| CSR | clinical study report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| DB | database |
| DBL | database lock |
| DBP | diastolic blood pressure |
| DRC | dosing review committee |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EMA | european medicines agency |





| Abbreviation | Definition |
|--------------|----------------------------------------------|
| eTMF | electronic trial master file |
| FDA | food and drug administration |
| HR | heart rate |
| IB | investigator's brochure |
| ICH | international council for harmonization |
| IWRS | interactive web-response system |
| LLOQ | lower limit of quantification |
| LOD | limit of detection |
| MedDRA | medical dictionary for regulatory activities |
| mITT | modified intent-to-treat population |
| NA | not applicable |
| NCS | non-clinically significant |
| PD | Parkinson's Disease |
| PE | physical examination |
| PK | pharmacokinetic |
| PD | protocol deviation |
| SAE | serious adverse event |
| SAF | safety analysis population |
| SAP | statistical analysis plan |





| Abbreviation | Definition |
|--------------|-------------------------------------------|
| SAS® | a software system used for data analysis |
| SBP | systolic blood pressure |
| SD | standard deviation |
| SE | standard error |
| SOC | system organ class |
| SOP | standard operating procedure |
| TEAE | treatment-emergent adverse event |
| TMF | trial master file |
| ULOQ | upper limit of quantification |
| UPDRS | Unified Parkinson's Disease Rating Scale |
| WHO | world health organization |
| WHO-DD | world health organization drug dictionary |